CLINICAL TRIAL: NCT04915534
Title: Evaluation of Gender Specific Differences in Postoperative Sore Throat Following General Anaesthesia With Ambu® AuraGain™ Laryngeal Mask
Brief Title: Gender Specific Differences in Postoperative Sore Throat for Ambu® AuraGain™ Laryngeal Mask
Acronym: LadyLAMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Katharina Epp, Dr.med. Katharina Epp, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 13715
Record Dates: First submitted 2021-05-21; First posted 2021-06-07 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Complications; Postoperative Pain
Keywords: postoperative sore throat and hoarseness (POST); laryngeal mask
MeSH Terms: conditions — Postoperative Complications; Pain, Postoperative; Hoarseness

STUDY DESIGN:
Intervention Model Description: prospective, randomized, controlled, single-blinded
Who Masked: Participant
Masking Description: Patients are allocated to the cuff pressure groups via block randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Women - low cuff pressure (Other): A cuff pressure of 45 cm H2O is used to block the laryngeal mask
  Interventions: Device: Ambu® AuraGain™ Laryngeal Mask (LM)
- Men - low cuff pressure (Other): A cuff pressure of 45 cm H2O is used to block the laryngeal mask
  Interventions: Device: Ambu® AuraGain™ Laryngeal Mask (LM)
- Women - normal cuff pressure (Other): A cuff pressure of 60 cm H2O is used to block the laryngeal mask
  Interventions: Device: Ambu® AuraGain™ Laryngeal Mask (LM)
- Men - normal cuff pressure (Other): A cuff pressure of 60 cm H2O is used to block the laryngeal mask
  Interventions: Device: Ambu® AuraGain™ Laryngeal Mask (LM)

INTERVENTIONS:
Device: Ambu® AuraGain™ Laryngeal Mask (LM) — Depending on the gender and randomization, the LM is either blocked with 45 cmH2O or with 60 cmH2O cuff pressure. Following general anaesthesia, patients are questioned for postop complications, with focus on postoperative sore throat and hoarseness.
  Other Names: Cuff pressure

SUMMARY:
The purpose of this study is to evaluate gender specific risk factors and the influence of cuff pressure in the occurrence of postoperative sore throat and hoarseness following general anaesthesia using Ambu® AuraGain™ Laryngeal Mask.

DETAILED DESCRIPTION:
The history and physical examinations of all patients scheduled for surgery are screened preoperatively for exclusion criteria. Patient recruitment is conducted by one of the study physicians. After eligibility is confirmed and written informed consent is obtained, enrolled participants are randomized depending on their gender (400 men, 400 women) in a single-blinded manner (patients) 24 hours before the intervention in a 1:1 ratio to low cuff pressure (45 cmH2O) or normal cuff pressure (60 cmH2O). Patient questioning via questionnaire is conducted in postoperative anaesthetic care unit, 24h, 48h and 72h until freedom of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery in ophthalmology under general anaesthesia with laryngeal mask
* Age > 18
* informed written consent

Exclusion Criteria:

* Anticipated difficult airway with indication for awake tracheal intubation
* Indication for RSI or elevated risk for aspiration;
* Pregnant or breastfeeding;
* Age < 18 years;
* Obesity
* Out-patient surgery (Geb. 505);
* Limited mouth opening;
* Pre-existing hoarseness and sore throat
* Participant in other studies
* Unable to provide informed written consent or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological gender (gender specific physiology of the Larynx)
Enrollment: 814 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Gender specific differences in sore throat 24 hours postoperative | 24 hours after general anaesthesia (removal of laryngeal mask)
  Comparing the incidence of postoperative sore throat between males and females within the first 24 hours after general anaesthesia with a second-generation Ambu® AuraGain™ Laryngeal Mask for elective, ophthalmological surgery
Differences in sore throat 24 hours postoperatively in correlation to cuff pressure | 24 hours after general anaesthesia (removal of laryngeal mask)
  Comparing the incidence of postoperative sore throat within the first 24 hours after general anaesthesia with a second-generation Ambu® AuraGain™ Laryngeal Mask for elective, ophthalmological surgery in correlation to cuff pressure (45 cmH2O and 60 cmH2O)

SECONDARY OUTCOMES:
Risk factors for postoperative sore throat in correlation to gender and cuff pressure | From end of general anaesthesia (removal of laryngeal mask) until at minimum Day 3. If symptoms persist past Day 3 postoperatively, the maximum observation period is 100 days or until freedom of symptoms (whichever comes first)
  Evaluating the effect of cuff pressure (45 cmH2O vs 60 cmH2O) stratified by gender on the incidence of postoperative sore throat (%). Furthermore, incidence of postoperative sore throat and hoarseness in PACU, at 48 and 72 hours until freedom of symptoms in correlation to gender and cuff pressure. In addition, influence of gender and cuff pressure on duration of pain and pain quality (measured via a pain scale of 0 = no pain, 1 = less than a cold, 2 = like a cold, 3 = more than a cold) will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology, University Medical Center of the Johannes Gutenberg-University, Mainz, Rhineland-Palatine, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaensson M, Gupta A, Nilsson U. Gender differences in sore throat and hoarseness following endotracheal tube or laryngeal mask airway: a prospective study. BMC Anesthesiol. 2014 Jul 19;14:56. doi: 10.1186/1471-2253-14-56. eCollection 2014. PMID 25061426
- [Derived] Epp K, Przybylski U, Luz C, Kriege M, Wittenmeier E, Schmidtmann I, Pirlich N. Evaluation of gender differences in postoperative sore throat and hoarseness following the use of Ambu AuraGain laryngeal mask: the randomised controlled LadyLAMA trial study protocol. BMJ Open. 2022 Jan 31;12(1):e056465. doi: 10.1136/bmjopen-2021-056465. PMID 35105650